CLINICAL TRIAL: NCT01680172
Title: Oral Ketamine in the Treatment of Depression and Anxiety in Patients With Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert P. Bright, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12-001156
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Cancer; Depression; Anxiety
Keywords: cancer; depression; anxiety; palliative care
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Single dose of ketamine (0.5 mg/kg)
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Single dose (0.5 mg/kg) of liquid ketamine 10mg/mL solution taken by mouth
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Single dose of liquid placebo solution taken by mouth
  Arms: Placebo

SUMMARY:
Depression is common in patients with cancer. Current medications for depression, while effective, take several weeks to take effect. Ketamine has emerged as a drug with promise for cancer patients. In two reported cases, a single dose of ketamine induced rapid and moderately sustained symptom reduction in depression and anxiety with no adverse side effects. Benefit was seen in as little as 1 hour and sustained up to 30 days. This study is a randomized, double-blind, placebo-controlled investigation testing whether a single dose of ketamine improves depression and anxiety relative to placebo in patients with cancer.

DETAILED DESCRIPTION:
Depression is common in patients with cancer. Current antidepressants, while effective, have an onset of action of at least several weeks. Ketamine has emerged as a drug with promise for cancer patients. It has been shown to potentiate opiate analgesic effects. Single dose parenteral and enteral administration studies in medically healthy treatment-resistant depressed patients have shown rapid relief of symptoms. A recent two patient case series reported a rapid and moderately sustained symptom reduction in depression and anxiety in palliative care patients following a single dose of oral ketamine 0.5 mg/kg, with no adverse effects. Benefit was seen as little as 1 hour after the administration and sustained up to 30 days. These case reports generate hypotheses of efficacy for ketamine in the treatment of depression and anxiety in patients with cancer. This study is a randomized, double-blind, placebo-controlled investigation of these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer
* Outpatient status at the time of study entry
* 18 years of age or older
* Life expectancy of at least 1 month
* Regular access to a telephone (for safety reasons)
* Reliable transportation to follow-up visits
* Caregiver observation available for 24 hours after the dose
* Histologically-proven malignancy
* Depression score of >11 on the Hospital Anxiety and Depression Scale (HADS)
* Provision of informed consent
* Able to complete the patient questionnaires alone or with assistance
* Able to speak and read English
* May receive other psycho-active medications while on the study i.e. opiates, except as defined within the exclusion criteria
* May receive psychotherapy from an outside provider at the beginning and/or during the course of the study

Exclusion Criteria:

* Obvious cognitive dysfunction or Mini Mental Status Exam score <20
* Antidepressants started or dose changed within 8 weeks of the beginning of the study or during the study
* Benzodiazepines prescribed for psychiatric indications that have been started or dose change within 2 weeks of the beginning of study enrollment
* Suicidal ideation or a suicide attempt within the last year
* Patients with current or past psychosis not from delirium
* Females who are pregnant or nursing
* Unable to take oral medications
* Primary or metastatic brain malignancy
* Gastrointestinal tract obstruction
* Prior adverse reaction to or other contraindication to ketamine
* Substance abuse or dependence, as defined by Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria, within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Bright, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Mayo Clinic in Scottsdale, Arizona from 2012 to 2014.
Groups:
- Ketamine: Single dose of ketamine (0.5 mg/kg)
  Ketamine: Single dose of ketamine (0.5 mg/kg)
- Placebo: Single dose of placebo
  Placebo: Single dose of placebo
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale - Anxiety Score (HADS-A)
Description: Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported in the literature to be >10 for anxiety and >8 for depression.
Time Frame: Baseline, 120 minutes
Population: Study was terminated early due to slow accrual.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 3 | 2
units on a scale
  HADS-A score at baseline | 12.3 (2.5) | 16.5 (4.9)
  HADS-A Score at 120 minutes post dose | 7.7 (3.8) | 11.0 (5.7)

2. Primary Outcome: Hospital Anxiety Depression Scale- Depression Score (HADS-D)
Description: as for outcome 1
Time Frame: Baseline, 120 minutes
Population: Study was terminated early due to slow accrual.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 3 | 2
units on a scale
  HADS-D Score at baseline | 12.7 (1.5) | 14.5 (2.1)
  HADS-D Score 120 minutes post dose | 11.7 (2.3) | 10.5 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated at baseline, 60 minutes and 120 minutes after study drug administration and Days 2, 7, 14 and 28 after study drug administration.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=3) | Placebo (N=2)
Rapid Heart Rate (Cardiac disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 2 (2) | 1 (1)
Impaired Concentration (General disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Drowsiness (General disorders) | 2 (2) | 2 (2)
Dizziness (General disorders) | 1 (1) | 1 (1)
Lightheaded (General disorders) | 1 (1) | 1 (1)
Confusion (General disorders) | 1 (1) | 1 (1)
Disorientation (General disorders) | 1 (1) | 1 (1)
Feeling high (General disorders) | 1 (1) | 0 (0)
Feeling of floating (General disorders) | 1 (1) | 0 (0)
Tingling sensation on skin (Nervous system disorders) | 1 (1) | 1 (1)
Impaired judgement (Psychiatric disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to slow accrual rate. Data analysis limited to 5 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes